CLINICAL TRIAL: NCT00691379
Title: Weekly Paclitaxel-carboplatin Plus Bevacizumab as First Line Therapy for Patients With Triple Negative (ER-,PR-,HER2-) Metastatic Breast Cancer. A Multicenter Phase I-II Study
Brief Title: Weekly Paclitaxel/Carboplatin/Bevacizumab as First Line Therapy for Triple Negative Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: Principal Investigator, VASSILIKI SXOINA, Prof. D. Mavroudis, Hellenic Oncology Research Group
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/08.02
Record Dates: First submitted 2008-05-29; First posted 2008-06-05 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Triple negative; Chemotherapy; Anti-angiogenesis therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Carboplatin; Bevacizumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Paclitaxel/Carboplatin/Bevacizumab
  Interventions: Drug: Carboplatin; Drug: Bevacizumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Carboplatin — Carboplatin (IV) 2 AUC on day 1,8,15. Treatment repeats every 4 weeks until progression
Drug: Bevacizumab — Bevacizumab (IV) 10 mg/kg on day 1,15. Treatment repeats every 4 weeks until progression
  Other Names: Avastin
Drug: Paclitaxel — Paclitaxel (IV) 90 mg/m2,on day 1,8,15. Treatment repeats every 4 weeks until progression
  Other Names: Taxoprol; Paxene; Taxol

SUMMARY:
This study will evaluate the efficacy of weekly paclitaxel-carboplatin combination plus bevacizumab as first line treatment in patients with metastatic triple negative breast cancer. Furthermore, the efficacy of the combination therapy will be correlated with the presence of circulating tumor cells (CTCs) in this population

DETAILED DESCRIPTION:
Breast cancer with absent or low expression of hormone receptors and HER2 (triple negative) does not respond to hormonal or biological therapy with trastuzumab. However, triple negative breast cancers are highly sensitive to chemotherapy. The combination of paclitaxel and carboplatin administered on a weekly basis is active and well tolerated. Recently, initial therapy of metastatic breast cancer with paclitaxel plus bevacizumab demonstrated prolonged progression-free survival, as compared with paclitaxel alone

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic breast adenocarcinoma
* No HER2 overexpression or gene amplification
* Absent or low ER or PR expression
* No previous therapy for metastatic breast cancer is allowed
* Age 18-75 years
* Measurable disease as defined by the presence of at least one measurable lesion (except bone metastases, ascites or pleural effusions)
* Performance status (WHO) 0-2
* Adequate liver (serum bilirubin <1.5 times the upper normal limit, AST and ALT <2.5 times the upper normal limit in the absence of demonstrable liver metastases, or <5 times the upper normal limit in the presence of liver metastases)
* adequate renal function (serum creatinine <1.5 times the upper normal limit)
* bone marrow (neutrophils ≥ 1.5x 109 /L, and platelets ≥ 100x 109 /L)
* No radiation of measurable disease (except brain metastases)
* No progressive brain metastases according to clinical or radiological criteria
* No brain metastases without prior radiation therapy
* Written informed consent

Exclusion Criteria:

* Active infection
* History of significant cardiac disease (unstable angina, congestive heart failure, myocardial infarction within the previous 6 months, ventricular arrhythmias)
* History of stroke
* Anticoagulation therapy (except of low dose aspirin <325mg)
* Other invasive malignancy except nonmelanoma skin cancer
* Psychiatric illness or social situation that would preclude study compliance
* Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | Objective responses confirmed by CT or MRI (on 3rd and 6th cycle)

SECONDARY OUTCOMES:
Toxicity profile | Toxicity assessment of each chemotherapy cycle
Time to Tumor Progression | 1-year
Overall Survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Mavrudis, MD, Principal Investigator — University Hospital of Crete
Locations (11):
- Greece (11):
  - University General Hospital of Alexandroupolis, Alexandroupoli
  - "IASO" General Hospital of Athens, 1st Dep of Medical Oncology, Athens
  - "Laikon" General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - "Marika Iliadis" Hospital of Athens, Dep of Medical Oncology, Athens
  - "Metaxa's" Anticancer Hospital of Piraeus, 1st Dep of Medical Oncology, Athens
  - 401 Military Hospital of Athens, Athens
  - Air Forces Military Hospital of Athens, Athens
  - University Hospital of Crete, Heraklion
  - State General Hospital of Larissa, Dep of Medical Oncology, Larissa
  - "Diabalkaniko" hospital, Thessaloniki, Thessaloniki
  - : "Theagenion" Anticancer Hospital of Thessaloniki, 2nd Dep of Medical Oncology, Thessaloniki

REFERENCES:
- [Derived] Saloustros E, Nikolaou M, Kalbakis K, Polyzos A, Christofillakis C, Kentepozidis N, Pistamaltzian N, Kourousis C, Vamvakas L, Georgoulias V, Mavroudis D. Weekly Paclitaxel and Carboplatin Plus Bevacizumab as First-Line Treatment of Metastatic Triple-Negative Breast Cancer. A Multicenter Phase II Trial by the Hellenic Oncology Research Group. Clin Breast Cancer. 2018 Feb;18(1):88-94. doi: 10.1016/j.clbc.2017.10.013. Epub 2017 Oct 24. PMID 29153775